CLINICAL TRIAL: NCT07160387
Title: Role of Gastrointestinal Endoscopy in Evaluation of Pediatric Failure to Thrive
Brief Title: Role of Gastroinestinal Endoscopy in Pediatric Failure to Thrive
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Abdelrady Abdelmalek, resident pediatric, Assiut University
Other Study IDs: GIT endoscopy in children FTT
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Failure to Thrive; Endoscope
MeSH Terms: conditions — Failure to Thrive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate the diagnostic role of gastrointestinal endoscopy in children presenting with failure to thrive and its correlation with histopathology and other diagnostic modalities.

DETAILED DESCRIPTION:
Failure to thrive (FTT) is a common and concerning clinical presentation in pediatric practice, characterized by inadequate growth or the inability to maintain expected weight and height percentiles (1). By accepted definitions, FTT can be defined as weight-for-age below the 5th percentile, or a drop of two major percentile lines on a standardized growth chart (2). It is not a diagnosis but rather a descriptive term that reflects an underlying issue with inadequate energy intake, absorption, or utilization. The causes of FTT are broad and often multifactorial, ranging from nutritional deficiencies and feeding difficulties to chronic infections, metabolic disorders, and gastrointestinal (GI) diseases. Among these, GI causes are particularly important, as they may be subtle, chronic, and potentially reversible with early diagnosis and appropriate management (3).

Despite advances in nutritional support and non-invasive diagnostics, a subset of children with persistent FTT require further evaluation to identify underlying organic causes (4). Gastrointestinal endoscopy, including esophagogastroduodenoscopy (EGD) and colonoscopy, provides direct visualization, tissue sampling, and diagnosis of a wide spectrum of pathologies such as gastroesophageal reflux disease, eosinophilic esophagitis, celiac disease, inflammatory bowel disease, peptic ulcer disease, and malabsorptive disorders (5).

Children presenting with FTT and associated gastrointestinal symptoms such as persistent vomiting, chronic diarrhea, abdominal pain, dysphagia, feeding intolerance, or hematemesis are particularly likely to benefit from gastrointestinal endoscopy (6). Even in the absence of overt GI symptoms, some children with unexplained FTT may harbor asymptomatic or minimally symptomatic conditions detectable only through endoscopic and histologic examination. Furthermore, gastrointestinal endoscopy can also help to rule out serious pathologies and provide reassurance to caregivers, allowing clinicians to focus on non-organic or psychosocial contributors to FTT when appropriate (7).

Despite its clinical utility, the use of gastrointestinal endoscopy in evaluation of FTT must be carefully considered due to its invasive nature, the need for sedation or anesthesia, and potential complications (8). Therefore, patient selection and risk-benefit ratio assessment are crucial. The decision to perform gastrointestinal endoscopy is often guided by a combination of clinical findings, laboratory data, growth patterns, and failure to respond to initial nutritional interventions (9).

ELIGIBILITY:
Inclusion Criteria:

1. Age from 6 months to 18 years..
2. Both sexes.
3. Diagnosed with failure to thrive, defined as :

   Weight-for-age below the 5th percentile for sex/age or crossing downward by ≥2 major percentiles, confirmed on two measurements.
4. Clinical suspicion of an underlying gastrointestinal cause (e.g., chronic vomiting, chronic diarrhea either bloody or not, chronic abdominal pain and/or gastrointestinal bleeding
5. Parental/guardian consent for their siblings to share in the study

Exclusion Criteria:

1. Known chronic disease already causing failure to thrive (genetic, cardiac, renal, or endocrine disorders).
2. Contraindications to endoscopy or anesthesia (e.g. severe coagulopathy, unstable cardiopulmonary status).
3. Parental refusal to participate or consent for endoscopy

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: any child from6 months to 18 years and has unexplained failure to thrive failure to thrive means: Weight-for-age below the 5th percentile for sex/age or crossing downward by ≥2 major percentiles lines on a standardized growth chart confirmed on two measurements.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2027-03-20 (Estimated); Study Completion 2027-04-20 (Estimated)

PRIMARY OUTCOMES:
Role of Gastrointestinal Endoscopy in Evaluation of Pediatric Failure to Thrive | baseline
  evaluate the diagnostic role of gastrointestinal endoscopy in children presenting with failure to thrive and its correlation with histopathology and other diagnostic modalities.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Burayzat S, Odeh M, Altamimi E, Al-Dweik S, El Wahab K, Alanasweh M, Al-Khraisat M, Barqawi M. Eesophagogastroduodenoscopy in paediatrics: does abiding by the international guidelines lead to appropriate management? A cross-sectional study. BMJ Open. 2022 Sep 1;12(9):e061489. doi: 10.1136/bmjopen-2022-061489. PMID 36581988
- [Background] Ngo PD, Lightdale JR. Advances in Pediatric Endoscopy. Gastroenterol Clin North Am. 2024 Dec;53(4):539-555. doi: 10.1016/j.gtc.2024.08.010. Epub 2024 Sep 30. PMID 39489574
- [Background] Sidhu R, Turnbull D, Haboubi H, Leeds JS, Healey C, Hebbar S, Collins P, Jones W, Peerally MF, Brogden S, Neilson LJ, Nayar M, Gath J, Foulkes G, Trudgill NJ, Penman I. British Society of Gastroenterology guidelines on sedation in gastrointestinal endoscopy. Gut. 2024 Jan 5;73(2):219-245. doi: 10.1136/gutjnl-2023-330396. PMID 37816587
- [Background] Lawson NR, Angelo J, Chiou E, Glinton K, Dean A. Failure to Thrive, Metabolic Acidosis, and Diarrhea in a 7-Week-Old Infant. Pediatrics. 2024 Sep 1;154(3):e2023064240. doi: 10.1542/peds.2023-064240. PMID 39086356
- [Background] Amil-Dias J, Oliva S, Papadopoulou A, Thomson M, Gutierrez-Junquera C, Kalach N, Orel R, Auth MK, Nijenhuis-Hendriks D, Strisciuglio C, Bauraind O, Chong S, Ortega GD, Fernandez SF, Furman M, Garcia-Puig R, Gottrand F, Homan M, Huysentruyt K, Kostovski A, Otte S, Rea F, Roma E, Romano C, Tzivinikos C, Urbonas V, Velde SV, Zangen T, Zevit N. Diagnosis and management of eosinophilic esophagitis in children: An update from the European Society for Paediatric Gastroenterology, Hepatology and Nutrition (ESPGHAN). J Pediatr Gastroenterol Nutr. 2024 Aug;79(2):394-437. doi: 10.1002/jpn3.12188. Epub 2024 Jun 24. PMID 38923067
- [Background] McDonald CM, Reid EK, Pohl JF, Yuzyuk TK, Padula LM, Vavrina K, Altman K. Cystic fibrosis and fat malabsorption: Pathophysiology of the cystic fibrosis gastrointestinal tract and the impact of highly effective CFTR modulator therapy. Nutr Clin Pract. 2024 Apr;39 Suppl 1:S57-S77. doi: 10.1002/ncp.11122. PMID 38429959
- [Background] Smith AE, Shah M, Badireddy M. Failure to Thrive. 2023 Nov 12. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK459287/ PMID 29083644
- [Background] Lin YC, Yen HR, Tsai FJ, Wang CH, Chien LC, Chen AC, Lin RT. Effects of cyproheptadine on body weight gain in children with nonorganic failure to thrive in Taiwan: A hospital-based retrospective study. PLoS One. 2021 Oct 19;16(10):e0258731. doi: 10.1371/journal.pone.0258731. eCollection 2021. PMID 34665812
- See also: Endoscopic biopsies - The gastrointestinal undercover agent! — https://journals.lww.com/jdap/fulltext/2025/01000/endoscopic_biopsies___the_gastrointestinal.2.aspx
- See also: Weight-Faltering in Infants and Children (Failure to Thrive) — https://ohiostate.elsevierpure.com/en/publications/weight-faltering-in-infants-and-children-failure-to-thrive